CLINICAL TRIAL: NCT03571568
Title: Phase 1/2a Trial of BI-1206, a Monoclonal Antibody to CD32b (FcyRIIB), in Combination With Rituximab With or Without Acalabrutinib in Subjects With Indolent B-Cell Non-Hodgkin Lymphoma That Has Relapsed or is Refractory to Rituximab
Brief Title: A Study of BI-1206 in Combination With Rituximab With or Without Acalabrutinib in Subjects With Indolent B-Cell NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-BI-1206-02
Record Dates: First submitted 2018-05-17; First posted 2018-06-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Indolent B-Cell Non-Hodgkin Lymphoma
MeSH Terms: interventions — Rituximab; acalabrutinib

STUDY DESIGN:
Intervention Model Description: Phase 1/2a, dose escalation, consecutive-cohort, open-label study trial of BI-1206 in combination with rituximab with or without Acalabrutinib
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- BI-1206 IV Dose Escalation (Experimental): Standard 3+3 Dose-Escalation of BI-1206 IV in combination with Rituximab
  Interventions: Biological: BI-1206; Biological: Rituximab
- BI-1206 SC Dose Escalation (Experimental): Adaptive Dose Escalation of BI-1206 SC (Bayesian logistic regression model (BLRM) in combination with Rituximab
  Interventions: Biological: BI-1206; Biological: Rituximab
- Phase 2a IV Dose expansion (Experimental): BI-1206 IV in Combination with Rituximab
  Interventions: Biological: BI-1206; Biological: Rituximab
- Phase 2a SC Signal seeking (Experimental): SC Arm, BI-1206 in Combination with Rituximab and Acalabrutinib
  Interventions: Biological: BI-1206; Biological: Rituximab; Biological: Acalabrutinib
- Phase 2a IV Signal Seeking (Experimental): IV Arm, BI-1206 in Combination with Rituximab and Acalabrutinib
  Interventions: Biological: BI-1206; Biological: Rituximab; Biological: Acalabrutinib

INTERVENTIONS:
Biological: BI-1206 — BI-1206 150 mg / 225 mg Subcutaneous injection
  BI-1206 50 mg /100 mg Intravenous infusion
Biological: Rituximab — Rituximab 375 mg/m2, as per SmPC
  Other Names: Ruxience
Biological: Acalabrutinib — Acalabrutinib 100 mg orally as per SmPC
  Other Names: Calquence
  Arms: Phase 2a IV Signal Seeking; Phase 2a SC Signal seeking

SUMMARY:
Phase 1/2a Clinical Trial of BI-1206, a Monoclonal Antibody to CD32b (FcyRIIB), in Combination with Rituximab with or without Acalabrutinib in Subjects with Indolent B-Cell Non-Hodgkin Lymphoma That has Relapsed or is Refractory to Rituximab

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter, dose escalation, consecutive-cohort, open-label trial of BI-1206 in combination with rituximab with or without acalabrutinib in subjects with indolent relapsed or refractory B-cell NHL, sub-types FL (except FL grade 3B), MZL, and MCL.

Phase 2a, consists of signal seeking cohorts followed by a randomized, parallel, two-arm dose optimization.

The trial consists of 2 main parts:

Phase 1

- Dose Escalation, with two different Arms assessing IV or SC dosing of BI-1206 in combination with rituximab, with dose escalation cohorts and selection of the IV and SC doses of BI-1206 for Phase 2a

Phase 2a

* Dose Expansion, with one expansion cohort evaluating the selected IV dose of BI-1206 in combination with rituximab
* Signal Seeking, assessing IV and SC dosing of BI-1206 in combination with rituximab and acalabrutinib. The Signal Seeking will consist of a Safety Run-in and an Expansion
* Dose Optimization to select the recommended dose of BI-1206 in combination with rituximab and acalabrutinib

ELIGIBILITY:
Inclusion Criteria:

1. Are ≥ 18 years of age by initiation of study treatment.
2. Have B-cell NHL proven by histology, with histological subtypes limited to follicular lymphoma (FL) (except FL grade 3B), MCL and marginal zone lymphoma (MZL)
3. Have measurable nodal disease
4. Are willing to undergo lymph node biopsies or biopsies of other involved tissue
5. Have relapsed disease or disease refractory to conventional treatment or for which no standard therapy exists
6. Have received at least one line of conventional previous therapy which must include at least one rituximab-based regimen
7. Have a life expectancy of at least 12 weeks
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
9. Have CD20+ malignancy
10. Have hematological and biochemical indices within prespecified ranges

Exclusion Criteria:

1. Have had an allogenic bone marrow or stem cell transplant within 12 months
2. Have presence of active chronic graft versus host disease
3. Have current leptomeningeal lymphoma or compromise of the central nervous system
4. Have transformed lymphoma from a pre-existing indolent lymphoma
5. Have Waldenstrom's Macroglobulinemia or FL grade 3B,
6. Need systemic doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) while on the study trial other than as pre-medication.
7. Have known or suspected hypersensitivity to rituximab or BI-1206
8. Have cardiac or renal amyloid light-chain amyloidosis
9. Have received any of the following:

   1. Chemotherapy or small molecule products with 2 weeks of first dose of BI-1206
   2. Radiotherapy (except for focal symptomatic control of lymphadenopathy) within 4 weeks
   3. Immunotherapy within 8 weeks
   4. Previous lines of treatment containing BTK inhibitors for Subjects receiving BI-1206 in combination with rituximab and acalabrutinib
10. Have ongoing toxic manifestations of previous treatments.
11. Have the ability to become pregnant (or already pregnant or lactating/breastfeeding).
12. Have had major surgery from which the subject has not yet recovered.
13. Are at high medical risk because of non-malignant systemic disease including active infection on treatment with antibiotics, antifungals or antivirals.
14. Are serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
15. Have an active, known or suspected autoimmune disease.
16. Have concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA])
17. Have current malignancies of other types

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Documenting AEs and SAEs and determining causality in relation to BI-1206 and/or rituximab and/or acalabrutinib | During the 28-day treatment period on induction therapy
  Assess the safety and tolerability profile of BI-1206 when administered intravenously (IV) or subcutaneously (SC) in combination with rituximab or rituximab and acalabrutinib in subjects with relapsed or refractory B-cell non-Hodgkin lymphoma (NHL), subtypes follicular lymphoma (FL)(except FL grade 3B), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL). Assessment will be done according to National Cancer Institute (NCI-CTCAE) criteria v. 5.0.
Determining the MTD of BI-1206 at the same dose level experiencing a BI-1206 or Rituximab-related or possibly related dose-limiting toxicity (DLT) | During the 28-day treatment period on induction therapy
  Phase 1:
  Select the recommended Phase 2 dose (RP2D) by establishing the maximum tolerated dose (MTD) of BI-1206 given once weekly for 4 weeks, via IV infusion or SC injection in combination with rituximab.
Determine the recommended dose of BI-1206 in combination with rituximab and acalabrutinib | During the 28-day treatment period on induction therapy
  Phase 2a:
  Select the recommended dose of BI-1206 in combination with rituximab and acalabrutinib.

SECONDARY OUTCOMES:
Evaluation of PK parameters for BI-1206 | Up to 1 year
  PK parameters assessed will include AUC, Cmax, time to Cmax and t1/2 of BI-1206 when administered IV or SC
Evaluation of ADA (immunogenicity) response to BI-1206 | Up to 1 year
  Assess the incidence and titre of antidrug antibodies of BI-1206 in serum when administered IV or SC in combination with rituximab or rituximab and acalabrutinib.
Measurement of peripheral blood B-lymphocytes depletion | Up to 1 year
  Evaluate the effect of BI-1206 administered IV or SC in combination with rituximab or rituximab and acalabrutinib measuring B Lymphocytes CD19+ (absolute value) as part of hematology assessment to determine the level of peripheral blood B lymphocyte depletion.
Assessment of overall response rate (ORR) according to the response criteria for malignant lymphoma (Cheson, 2014). | Up to 1 year
  Assess possible anti-tumor activity of BI-1206 administered IV or SC in combination with rituximab or rituximab and acalabrutinib at Week 6 after first dose of BI-1206 and for subjects who continue during maintenance therapy.

OTHER OUTCOMES:
Expression levels of CD32b protein | Up to 1 year
  To investigate CD32b protein expression levels using flow cytometry to evaluate any potential correlation with clinical responses. Change from baseline expression levels will be summarized descriptively by dose cohort and/or response to treatment.
Assessment of Patient Reported Outcomes using the NCI PRO-CTCAE questionnaire | Up to 1 year
  The NCI PRO-CTCAE will be used to evaluate symptomatic toxicities reported by patients. The questionnaire characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities, all toxicities that can be meaningfully reported from the patient perspective.
  Responses are scored from 0 to 4 (or 0/1 for absent/present). Scores for each attribute (frequency, severity and/or interference) will be presented descriptively (e.g. summary statistics or graphical presentations).
Expression levels of CD32b and/or other immunological markers | Up to 1 year
  Perform whole-transcriptome, quantitative polymerase chain reaction (qPCR) and/or IHC analysis of lymph node biopsies to evaluate potential correlation with clinical responses.
Measurement of serum cytokines levels and/or soluble CD32b. | Up to 1 year
  Study the potential cause of infusion related reactions (IRRs), such as cytokine release signs, C-reactive protein (CRP) and/or soluble CD32b.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Norton Cancer Institute - St. Matthews 3991 Dutchmans Lane Medical Plaza II, Suite 405, Louisville, Kentucky
- Brazil (10):
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - A.C. Camargo Cancer Center, São Paulo
  - Hospital Amaral Carvalho, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Samaritano, São Paulo
  - Hospital Sírio-Libanês, São Paulo
- Germany (2):
  - Krankenhaus Nordwest Klinik für Onkologie und Hämatologie, Frankfurt am Main, Hesse
  - Robert Bosch Hospital, Dep of Hematology, Oncology and Palliative care, Stuttgart
- Poland (2):
  - Szpital Specjlistyczny, Grudziądz
  - Małopolskie Centrum Medyczne, Krakow
- Spain (9):
  - Hospital ICO, Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Dep Hematologia, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Marañon-Oncología Médica, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - University Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital University Virgen Macarene, Seville
- Sweden (2):
  - Department of Oncology, Skåne University Hospital, Lund
  - Department of Oncology, Academical Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
All information concerning the product as well as any matter concerning the operation of the Sponsor, such as clinical indications for the drug, its formula, methods of manufacture and other scientific data relating to it, that have been provided by the Sponsor and are unpublished, are confidential and must remain the sole property of the Sponsor. The Investigator will agree to use the information only for the purposes of carrying out this study and for no other purpose unless prior written permission from the Sponsor is obtained.
Supporting Information: Study Protocol, CSR
Time Frame: Within one year from end of study
Access Criteria: Paper copy of CSR